CLINICAL TRIAL: NCT04158544
Title: Immune Monitoring During Systemic Therapy of Metastatic Malignant Melanoma
Brief Title: Immune Monitoring in Metastatic Melanoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Edward Geissler, Head of Experimental Surgery, University of Regensburg
Other Study IDs: 16-101-0125
Record Dates: First submitted 2019-10-23; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Melanoma
Keywords: Immune monitoring; Immunotherapy
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples (10ml EDTA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Checkpoint Inhibitors: Patients with metastatic melanoma receiving systemic therapy with checkpoint inhibitors
- Kinase Inhibitors: Patients with metastatic melanoma receiving systemic therapy with kinase inhibitors

SUMMARY:
The mean survival time in the advanced tumor stage in the presence of distant metastases in malignant melanoma was less than 9 months until a few years ago. Intensive research efforts have led to the development of promising new therapeutic strategies and their clinical application. These include on the one hand mutation-specific inhibitors of important for cell division serine-threonine kinase BRAF such as vemurafenib, dabrafenib and encorafenib and inhibitors of the downstream target protein, the mitogen-activated protein kinase kinase (MEK), such as trametinib, binimetinib and cobimetinib.

The group of immunotherapeutics is a second new class of drugs, in which great hope for the treatment of metastatic melanoma is placed. Antibody-mediated blockage of surface molecules expressed on immune cells, referred to as immune checkpoints, results in activation of the immune system. As a result, an anti-tumor immune response is triggered, which has led to considerable therapeutic success in metastatic melanoma. To date, three checkpoint inhibitors have been approved for the treatment of metastatic melanoma. Ipilimumab is an antibody that binds cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4); Pembrolizumab and nivolumab cause immune stimulation by binding the Programmed Death Receptor (PD1).

However, the impact of the therapy on the immune system as a whole is largely unknown. A comprehensive understanding of these effects is crucial to be able to further develop the therapy and to evaluate useful combination therapies with other immunomodulatory agents.

Within the framework of this project changes of the immune response under a systemic therapy of the malignant melanoma are to be characterized. The material for the analysis comes from blood samples collected during routine patient check-ups.

The aim of the analyzes is to precisely characterize the effects of the different therapeutics on the function of the immune system. In particular, the study will investigate whether certain therapeutic agents can weaken or activate the immune system and thus, in addition to the direct effect on the tumor cells, mediate indirect therapeutic effects via immune modulation. In the long term, the investigators want to use the knowledge gained to further improve the already existing therapeutic strategies of malignant melanoma by additional modulation of the immune system.

DETAILED DESCRIPTION:
Despite recent breakthroughs in the treatment of melanoma, the prognosis in the advanced stage of the disease continues to be very poor. 45-50% of all melanomas carry a point mutation in codon 600 of the BRAF gene encoding a serine-threonine kinase. The two most common BRAF mutations (V600E and V600K) constitutively activate the MAP kinase signaling pathway that drives the proliferation and survival of cancer cells. Specific BRAF V600 inhibitors such as vemurafenib, dabrafenib and encorafenib and inhibitors of the downstream target MEK such as trametinib, binimetinib and cobimetinib are very effective regimens in BRAF-positive metastatic melanoma.

Recent studies have shown that these inhibitors in addition to the effects on the tumor cells also have an influence on cells of the immune system. For example, vemurafenib leads to a loss of peripheral blood lymphocytes. Thus, the number of peripheral CD4 + positive cells decreases with vemurafenib therapy, while the number of natural killer cells (NK cells) increases. On the other hand, initial studies show that B cells and CD8 + positive cells are not affected numerically by vemurafenib. It has been demonstrated that vemurafenib but not dabrafenib reduces the number of peripheral lymphocytes in melanoma patients and changes the function and phenotype of CD4 + positive cells, although both drugs show comparable clinical efficacy. Selective inhibition of BRAF by inhibitors such as vemurafenib or dabrafenib thus has a significant influence on the peripheral lymphocyte populations of melanoma patients. Studies have been demonstrated that inhibition of BRAF can induce increased invasion of tumor-infiltrating lymphocytes into melanoma metastases. Tumor infiltration of CD4 + and CD8 + positive lymphocytes is surprisingly enhanced by therapy with a BRAF inhibitor. Furthermore, it could be shown in this study that the number of immunoreactive cells correlated with a reduction in tumor size and an increased necrosis in the tumor areas. The data obtained so far suggest that treatment with BRAF inhibitors increases melanoma antigen expression and thus facilitates T cell cytotoxicity. This results in a more favorable tumor microenvironment for a synergistic BRAF-targeted therapy and immunotherapy. This therapeutic strategy is currently being evaluated in clinical trials.

The group of immunotherapeutics is a second new class of drugs, in which great hope for the treatment of metastatic melanoma is placed. Ipilimumab is an antibody that binds the cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4), thereby stimulating T-cell activation and proliferation. The drug has been approved for the treatment of metastatic melanoma since July 2011 and significantly increases survival in some patients. In addition, at the end of 2015, a monoclonal antibody directed against the Programmed Death Receptor (PD1) was approved by the European Medicines Commission for the treatment of unresectable or metastatic melanoma. PD1 is a receptor that is expressed on T cells and inhibits T cell activation upon binding of a ligand. Study results have shown that blocking this T-cell inhibition with PD1 or PD-L1 antagonists is a very effective therapeutic strategy for melanoma and other tumor entities.

Current data show that targeted therapy has a major impact on the tumor microenvironment and on the regulatory and effector cells of the immune system. However, the impact of the therapy on the immune system as a whole is largely unknown. A comprehensive understanding of these effects is crucial to be able to further develop the therapy and to evaluate useful combination therapies with other immunomodulatory agents.

In the context of this study, the immune status, e.g. the number and the activation state of different immune cells at the beginning and in the course of a systemic therapy for metastatic melanoma should be determined. For this purpose, 10 ml of EDTA blood is taken as part of the guideline-compliant routine care (The blood samples taken in the study are given every 4 weeks for therapy with kinase inhibitors and every 2 weeks for therapy with checkpoint inhibitors). The blood samples taken before and during therapy will be analyzed by flow cytometry and the changes in the immunophenotype will be correlated with the response to therapy. In this way, the investigator want to identify both predictive and prognostic markers. The assessment of the immune status should help to optimize the effectiveness of melanoma therapy. Therefore, it would be important to identify suitable markers and to characterize subgroups of immune cells that have an impact on the tumor microenvironment.

The evaluation of the immune status in melanoma patients could thus be incorporated into the treatment strategies in the future in order to combine a targeted therapy with immunomodulating substances or also from enriched sub-populations of immune cells in order to increase the effectiveness of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Presence of metastatic melanoma expecting treatment with immune or targeted therapy

Exclusion Criteria:

* <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic melanoma of all ages and both sexes will be screened for inclusion if they qualify for systemic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in frequency of peripheral immune cell populations assessed by immune monitoring through flow cytometry (ONE study FACS panel) | Before start of treatment, 3 and 6 weeks after start of treatment as well as through study completion, an average of 1 year
  As part of the course of therapy during routine check-up, blood samples are collected and then analyzed by flow cytometry (ONE study panel). Frequency of surface antigens of PBMC are analyzed and the characterized sub-populations are monitored during the follow-up. Thereby, changes in frequency of surface antigens will be assessed compared to baseline (before start of treatment). This allows to determine the individual immunophenotype of a patient.
Change in activation status of peripheral immune cell populations assessed by immune monitoring through flow cytometry (ONE study FACS panel) | Before start of treatment, 3 and 6 weeks after start of treatment as well as through study completion, an average of 1 year
  As part of the course of therapy during routine check-up, blood samples are collected and then analyzed by flow cytometry (ONE study panel). Expression level of surface antigens of PBMC are analyzed and the characterized sub-populations are monitored during the follow-up. Thereby, changes in expression level of surface antigens will be assessed compared to baseline (before start of treatment). This allows to determine the individual immunophenotype of a patient.

SECONDARY OUTCOMES:
Liver inflammation (ALT) | Before start of treatment, 3 and 6 weeks after start of treatment as well as through study completion, an average of 1 year
  Screening for liver inflammation (serum ALT U/l)
Liver inflammation (AST) | Before start of treatment, 3 and 6 weeks after start of treatment as well as through study completion, an average of 1 year
  Screening for liver inflammation (serum AST U/l)

CONTACTS AND LOCATIONS:
Overall Officials: Edward K Geissler, Phd, Principal Investigator — Dept. of Exp. Surgery, University Hospital Regensburg
Locations (1):
- Dept. of Dermatology; Univeristy Hospital Regensburg, Regensburg, Bavaria, Germany

REFERENCES:
- [Background] Chapman PB, Hauschild A, Robert C, Haanen JB, Ascierto P, Larkin J, Dummer R, Garbe C, Testori A, Maio M, Hogg D, Lorigan P, Lebbe C, Jouary T, Schadendorf D, Ribas A, O'Day SJ, Sosman JA, Kirkwood JM, Eggermont AM, Dreno B, Nolop K, Li J, Nelson B, Hou J, Lee RJ, Flaherty KT, McArthur GA; BRIM-3 Study Group. Improved survival with vemurafenib in melanoma with BRAF V600E mutation. N Engl J Med. 2011 Jun 30;364(26):2507-16. doi: 10.1056/NEJMoa1103782. Epub 2011 Jun 5. PMID 21639808
- [Background] Board RE, Ellison G, Orr MC, Kemsley KR, McWalter G, Blockley LY, Dearden SP, Morris C, Ranson M, Cantarini MV, Dive C, Hughes A. Detection of BRAF mutations in the tumour and serum of patients enrolled in the AZD6244 (ARRY-142886) advanced melanoma phase II study. Br J Cancer. 2009 Nov 17;101(10):1724-30. doi: 10.1038/sj.bjc.6605371. Epub 2009 Oct 27. PMID 19861964
- [Background] Schilling B, Paschen A. Immunological consequences of selective BRAF inhibitors in malignant melanoma: Neutralization of myeloid-derived suppressor cells. Oncoimmunology. 2013 Aug 1;2(8):e25218. doi: 10.4161/onci.25218. Epub 2013 Jun 10. PMID 24167759
- [Background] Schilling B, Sucker A, Griewank K, Zhao F, Weide B, Gorgens A, Giebel B, Schadendorf D, Paschen A. Vemurafenib reverses immunosuppression by myeloid derived suppressor cells. Int J Cancer. 2013 Oct 1;133(7):1653-63. doi: 10.1002/ijc.28168. Epub 2013 Apr 13. PMID 23526263
- [Background] Schilling B, Sondermann W, Zhao F, Griewank KG, Livingstone E, Sucker A, Zelba H, Weide B, Trefzer U, Wilhelm T, Loquai C, Berking C, Hassel J, Kahler KC, Utikal J, Al Ghazal P, Gutzmer R, Goldinger SM, Zimmer L, Paschen A, Hillen U, Schadendorf D; DeCOG. Differential influence of vemurafenib and dabrafenib on patients' lymphocytes despite similar clinical efficacy in melanoma. Ann Oncol. 2014 Mar;25(3):747-753. doi: 10.1093/annonc/mdt587. Epub 2014 Feb 6. PMID 24504444
- [Background] Wilmott JS, Long GV, Howle JR, Haydu LE, Sharma RN, Thompson JF, Kefford RF, Hersey P, Scolyer RA. Selective BRAF inhibitors induce marked T-cell infiltration into human metastatic melanoma. Clin Cancer Res. 2012 Mar 1;18(5):1386-94. doi: 10.1158/1078-0432.CCR-11-2479. Epub 2011 Dec 12. PMID 22156613
- [Background] Frederick DT, Piris A, Cogdill AP, Cooper ZA, Lezcano C, Ferrone CR, Mitra D, Boni A, Newton LP, Liu C, Peng W, Sullivan RJ, Lawrence DP, Hodi FS, Overwijk WW, Lizee G, Murphy GF, Hwu P, Flaherty KT, Fisher DE, Wargo JA. BRAF inhibition is associated with enhanced melanoma antigen expression and a more favorable tumor microenvironment in patients with metastatic melanoma. Clin Cancer Res. 2013 Mar 1;19(5):1225-31. doi: 10.1158/1078-0432.CCR-12-1630. Epub 2013 Jan 10. PMID 23307859
- [Background] Robert C, Ribas A, Wolchok JD, Hodi FS, Hamid O, Kefford R, Weber JS, Joshua AM, Hwu WJ, Gangadhar TC, Patnaik A, Dronca R, Zarour H, Joseph RW, Boasberg P, Chmielowski B, Mateus C, Postow MA, Gergich K, Elassaiss-Schaap J, Li XN, Iannone R, Ebbinghaus SW, Kang SP, Daud A. Anti-programmed-death-receptor-1 treatment with pembrolizumab in ipilimumab-refractory advanced melanoma: a randomised dose-comparison cohort of a phase 1 trial. Lancet. 2014 Sep 20;384(9948):1109-17. doi: 10.1016/S0140-6736(14)60958-2. Epub 2014 Jul 15. PMID 25034862
- [Background] Merelli B, Massi D, Cattaneo L, Mandala M. Targeting the PD1/PD-L1 axis in melanoma: biological rationale, clinical challenges and opportunities. Crit Rev Oncol Hematol. 2014 Jan;89(1):140-65. doi: 10.1016/j.critrevonc.2013.08.002. Epub 2013 Aug 28. PMID 24029602
- [Background] Streitz M, Miloud T, Kapinsky M, Reed MR, Magari R, Geissler EK, Hutchinson JA, Vogt K, Schlickeiser S, Kverneland AH, Meisel C, Volk HD, Sawitzki B. Standardization of whole blood immune phenotype monitoring for clinical trials: panels and methods from the ONE study. Transplant Res. 2013 Oct 25;2(1):17. doi: 10.1186/2047-1440-2-17. PMID 24160259